CLINICAL TRIAL: NCT03794440
Title: A Randomized, Open-label，Multi-center Study to Evaluate the Efficacy and Safety of the Combination of Sintilimab and IBI305 Compared to Sorafenib in the First-Line Treatment of Patients With Advanced Hepatocellular Carcinoma. （ORIENT-32）
Brief Title: A Study to Evaluate the Efficacy and Safety of Sintilimab in Combination With IBI305 (Anti-VEGF Monoclonal Antibody) Compared to Sorafenib as the First-Line Treatment for Advanced Hepatocellular Carcinoma.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI338B301
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab +IBI305 (Experimental)
  Interventions: Drug: Sintilimab; Drug: IBI305
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sintilimab — 200mg IV d1， Q3W
  Other Names: IBI308
  Arms: Sintilimab +IBI305
Drug: IBI305 — 15mg/kg IV d1， Q3W
  Other Names: anti-VEGF monoclonal antibody
  Arms: Sintilimab +IBI305
Drug: Sorafenib — 400mg PO BID
  Arms: Sorafenib

SUMMARY:
The purpose of the study is to assess the safety, tolerability and effectiveness of Sintilimab in combination with IBI305 in patients with HCC as the first-line treatment compared with Sorafenib. This study is a randomised, Open-label，Multi-center Study. The primary endpoint is overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma confirmed by histology/cytology. Cirrhosis meets the clinical diagnostic criteria for hepatocellular carcinoma of the American Association for the Diagnosis of Liver Diseases (AASLD).
2. ECOG performance status between 0 and 1
3. No systematic anti-tumor treatment has been performed.(End of postoperative adjuvant chemotherapy for more than 6 months allowed).
4. Barcelona Clinic Liver Cancer stage C. BCLC stage B, not suitable for radical surgery and/or local treatment.
5. At least 1 lesion with measurable disease at baseline by RECIST V1.1.
6. Child-Pugh: <=7
7. Adequate organ and bone marrow function.

Exclusion Criteria:

1. With fibrous lamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma components in tumor tissues.
2. Have a history of hepatic encephalopathy or have a history of liver transplantation.
3. With clinical symptoms requires drainage of pleural effusion, ascites or pericardial effusion.
4. Central nervous system (CNS) metastasis.
5. Uncontrolled high blood pressure, systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg after optimal medical treatment.
6. Local treatment for liver lesions within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | up to 24 months after randomization
Progression-free survival (PFS) | up to 24 months after randomization
  Progression-free survival (PFS) in two arms based on RECIST V1.1 by Independent Radiological Review Committee, IRRC.

SECONDARY OUTCOMES:
PFS | up to 24 months after randomization
  PFS in two arms based on RECIST V1.1 by investigator.
Objective response rate (ORR) | up to 24 months after randomization
  Objective response rate (ORR) in two arms based on RECIST V1.1 by IRRC and investigator .
Disease control rate (DCR) | up to 24 months after randomization
  DCR in two arms based on RECIST V1.1 by IRRC and investigator.
Duration of response (DOR) | up to 24 months after randomization
  DOR in two arms based on RECIST V1.1 by IRRC and investigator.
Time to progression (TTP) | One assessment was performed every 6 weeks (±7 days) from the time of randomization, and once every 12 weeks (±7 days) after 48 weeks.
  TTP in two arms based on RECIST V1.1 by IRRC and investigator.
Time to response (TTR) | up to 24 months after randomization
  TTR in two arms based on RECIST V1.1 by IRRC and investigator.
PFS | up to 24 months after randomization
  PFS in two arms based on mRECIST by IRRC.
Objective response rate (ORR) | up to 24 months after randomization
  Objective response rate (ORR) in two arms based on mRECIST by IRRC.
Time to progression (TTP) | up to 24 months after randomization
  TTP in two arms based on mRECIST by IRRC.
Duration of response (DOR) | up to 24 months after randomization
  DOR in two arms based on mRECIST by IRRC.
Disease control rate (DCR) | up to 24 months after randomization
  DCR in two arms based on mRECIST by IRRC.
Time to response (TTR) | up to 24 months after randomization
  TTR in two arms based on mRECIST by IRRC.
Anti-drug antibody (ADA) | up to 24 months after randomization
  Immunogenicity measured by anti-drug antibody (ADA) for Sintilimab and IBI305.
EORTC QLQ-C30 | up to 24 months after randomization
EORTC QLQ-HCC18 | up to 24 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ren Z, Xu J, Bai Y, Xu A, Cang S, Du C, Li Q, Lu Y, Chen Y, Guo Y, Chen Z, Liu B, Jia W, Wu J, Wang J, Shao G, Zhang B, Shan Y, Meng Z, Wu J, Gu S, Yang W, Liu C, Shi X, Gao Z, Yin T, Cui J, Huang M, Xing B, Mao Y, Teng G, Qin Y, Wang J, Xia F, Yin G, Yang Y, Chen M, Wang Y, Zhou H, Fan J; ORIENT-32 study group. Sintilimab plus a bevacizumab biosimilar (IBI305) versus sorafenib in unresectable hepatocellular carcinoma (ORIENT-32): a randomised, open-label, phase 2-3 study. Lancet Oncol. 2021 Jul;22(7):977-990. doi: 10.1016/S1470-2045(21)00252-7. Epub 2021 Jun 15. PMID 34143971